CLINICAL TRIAL: NCT06524232
Title: The STop UNhealthy Substance Use Now Trial
Acronym: STUN II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Ohio Association of Community Health Centers (OACHC) (Unknown); Bon Secours Mercy Health (BSMH) (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dan.Jonas, Director and Professor, Division of General Internal Medicine, Ohio State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R18HS029782-01 (AHRQ)
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Risky Health Behavior; Substance Use Disorders; Substance Abuse; Alcohol Use Disorder; Drinking, Alcohol; Substance Use
MeSH Terms: conditions — Health Risk Behaviors; Substance-Related Disorders; Alcoholism; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: STUN II is a 48-site randomized 2x2 factorial trial to evaluate the comparative effectiveness of implementation strategies, including practice facilitation (PF), PF + learning collaborative (LC), PF + performance incentives (PI), and PF+LC+PI, on implementation of screening for and delivery of evidence-based interventions for substance use disorders (SUD) in primary care. We will use a stratified block randomization strategy with a block size of 12 practices to ensure a high degree of balance between study arms. The implementation phase will last for 12 months, and we will conduct 12-month post-implementation assessments to assess sustainment. The 2x2 design will allow us to assess the improvement in rates of screening and delivery of evidence-based interventions for SUDs in primary care with PF alone and the incremental benefit of LC, PI, or their combination, to inform primary care practices and health systems about optimal implementation strategies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Practice Facilitation Only (Active Comparator): Practice Facilitation: Practices will receive up to 2 hours of direct practice facilitation services per month for 12 months.
  Interventions: Other: Practice Facilitation (PF)
- Practice Facilitation + Learning Collaborative (Experimental): Practice Facilitation (PF): Practices will receive up to 2 hours of direct practice facilitation services per month for 12 months.
  Learning Collaborative (LC): Virtual LC sessions will be held monthly and will include participants presenting anonymized cases to clinical experts, targeted brief didactics related to the content of the cases, and time for open discussion and Q&A.
  Interventions: Other: Practice Facilitation (PF); Other: Learning Collaborative (LC)
- Practice Facilitation + Performance Incentives (Experimental): Practice Facilitation: Practices will receive up to 2 hours of direct practice facilitation services per month for 12 months.
  Performance Incentives: Practices will receive a maximum total of $6,000 based on their performance during the 12-month implementation period. They will have the opportunity to receive up to $1,500 per quarter if they reach performance milestones for the quarter.
  Interventions: Other: Practice Facilitation (PF); Other: Performance Incentives (PI)
- Practice Facilitation + Learning Collaborative + Performance Incentives (Experimental): Practice Facilitation: Practices will receive up to 2 hours of direct practice facilitation services per month for 12 months.
  Learning Collaborative (LC): Virtual LC sessions will be held monthly and will include participants presenting anonymized cases to clinical experts, targeted brief didactics related to the content of the cases, and time for open discussion and Q&A.
  Performance Incentives: Practices will receive a maximum total of $6,000 based on their performance during the 12-month implementation period. They will have the opportunity to receive up to $1,500 per quarter if they reach performance milestones for the quarter.
  Interventions: Other: Practice Facilitation (PF); Other: Learning Collaborative (LC); Other: Performance Incentives (PI)

INTERVENTIONS:
Other: Practice Facilitation (PF) — Practices will meet with practice facilitators monthly and apply tests of change using a Plan-Do-Study-Act approach, guided by the PF team. Facilitators will confirm that practices have established workflows for substance use disorder (SUD) screening and interventions and perform checks periodically to ensure progression. PF will entail: implementing protocols/algorithms for evidence-based screening and interventions, promoting decision support tools and templates to support practice workflow, optimizing electronic health record (EHR) use to pull clinical data monthly to guide the improvement process, developing patient registries (e.g., for those with SUD) to identify needed care and optimize delivery of evidence-based interventions, encouraging proactive, team-based care with assigned roles and responsibilities, and enhancing the understanding of evidence-based SUD interventions, including counseling and referral resources to ensure practices have appropriate intervention options.
Other: Learning Collaborative (LC) — Virtual LC sessions will be held monthly and will include participants presenting anonymized cases to clinical experts, targeted brief didactics related to the content of the cases, and time for open discussion and Q&A. Participant-generated ideas for topics to be covered during virtual LC sessions will be encouraged. Some specific topics will include optimal SUD screening approaches; prescribing medications for opioid use disorder (OUD) in primary care; pragmatic issues around integrated SUD care within primary care such as compliance with state and federal requirements, note templates/visit frequency, and when/how to escalate care for patients with severe or worsening SUD; medications for alcohol use disorder (AUD); and motivational interviewing.
  Arms: Practice Facilitation + Learning Collaborative; Practice Facilitation + Learning Collaborative + Performance Incentives
Other: Performance Incentives (PI) — We will work closely with key stakeholders and the Steering Committee to co-design the PI strategy, refining the specific performance metrics to ensure that they align with other ongoing efforts in our partnering organizations. We plan to base the incentive on achieving a threshold target for the percentage of eligible adult patients screened for SUD, or the percentage improvement in screening, for quarters 1 and 2. For quarters 3 and 4, after practices have had time to implement and improve their processes for screening for SUD, the incentives will evolve to become a composite of (1) patients screened for SUD (the same as used in quarters 1 and 2) and (2) achieving a threshold target for the percentage of persons with SUD who received evidence-based interventions.
  Arms: Practice Facilitation + Learning Collaborative + Performance Incentives; Practice Facilitation + Performance Incentives

SUMMARY:
The STop UNhealthy (STUN) Substance Use Now Trial (STUN II) is a multisite trial aiming to evaluate the comparative effectiveness of the following strategies for improving the implementation of screening and interventions for substance use disorders in primary care: practice facilitation (PF), PF plus a learning collaborative (LC), PF plus performance incentives (PI), and PF+LC+PI. We plan to enroll 144 clinic staff participants from 48 primary care practices

DETAILED DESCRIPTION:
The STop UNhealthy (STUN) Substance Use Now Trial (STUN II) is a multisite trial aiming to evaluate the comparative effectiveness of the following strategies for improving the implementation of screening and interventions for substance use disorders in primary care: practice facilitation (PF), PF plus a learning collaborative (LC), PF plus performance incentives (PI), and PF+LC+PI. We plan to enroll 144 clinic staff participants from 48 primary care practices

Specific aim 1 (primary aim) will compare the effect of learning collaborative (LC) participation, performance incentives (PI), or their combination, with practice facilitation (PF) only, on implementation of evidence-based screening for SUDs.

Specific aim 2 (secondary aim) will compare the effect of LC participation, PI, or their combination, with PF only, on implementation of evidence-based interventions for SUDs, including (a) brief counseling, (b) medications (e.g., buprenorphine, naltrexone) and adherence to them, and (c) referral to specialty care.

Specific aims 1 and 2 will produce fundamentally important evidence about the comparative effectiveness of PF, PF+LC, PF+PI, and PF+LC+PI strategies on uptake of evidence-based screening and interventions for SUD when delivered to primary care practices.

Specific aim 3 (exploratory aim) will use a longitudinal mixed-methods evaluation to assess the association between implementation effectiveness and putative moderators (e.g., organizational readiness for change) and mediators (e.g., implementation climate). Aim 3 will generate scientific knowledge about mechanisms of change (why and how the various strategies work) in primary care settings.

ELIGIBILITY:
Inclusion Criteria:

* Clinic staff members from primary care practices who provide care for adult patients and have a leadership role within the practice (e.g. lead physician, practice manager, lead medical assistant/nurse, clinical champion)

Exclusion Criteria:

* Clinic staff members who already have ongoing involvement in programs that would conflict with or preclude this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of adults screened for substance use disorder | 12 months
  Number of people aged 18 and older who are screened for substance use disorder using a validated screening tool
Percent of adults screened for substance use disorder | 12 months
  Percent of people aged 18 and older who are screened for substance use disorder using a validated screening tool

SECONDARY OUTCOMES:
Number of adults with a positive screen for substance use disorder | 12 months
  Of those aged 18 and older who were screened for substance use disorder, number who had a positive screening result
Number of adults with a positive screen for substance use disorder | 24 months
  Of those aged 18 and older who were screened for substance use disorder, number who had a positive screening result
Percent of adults with a positive screen for substance use disorder | 12 months
  Of those aged 18 and older who were screened for substance use disorder, percentage who had a positive screening result
Percent of adults with a positive screen for substance use disorder | 24 months
  Of those aged 18 and older who were screened for substance use disorder, percentage who had a positive screening result
Number of adults who received any evidence-based intervention for substance use disorder | 12 months
  Of those aged 18 or older who were identified as having substance use disorder and/or alcohol use disorder, number who received brief counseling, medication, or referral to specialty care
Number of adults who received any evidence-based intervention for substance use disorder | 24 months
  Of those aged 18 or older who were identified as having substance use disorder and/or alcohol use disorder, number who received brief counseling, medication, or referral to specialty care
Percentage of adults who received any evidence-based intervention for substance use disorder | 24 months
  Of those aged 18 or older who were identified as having substance use disorder and/or alcohol use disorder, percentage that received brief counseling, medication, or referral to specialty care
Percentage of adults who received any evidence-based intervention for substance use disorder | 12 months
  Of those aged 18 or older who were identified as having substance use disorder and/or alcohol use disorder, percentage that received brief counseling, medication, or referral to specialty care
Number of adults who received brief counseling for substance use disorder | 12 months
  Of people aged 18 or older who screened positive for substance use disorder and/or alcohol use disorder, number who received brief counseling
Number of adults who received brief counseling for substance use disorder | 24 months
  Of people aged 18 or older who screened positive for substance use disorder and/or alcohol use disorder, number who received brief counseling
Percentage of adults who received brief counseling for substance use disorder | 24 months
  Of people aged 18 or older who screened positive for substance use disorder and/or alcohol use disorder, percentage who received brief counseling
Percentage of adults who received brief counseling for substance use disorder | 12 months
  Of people aged 18 or older who screened positive for substance use disorder and/or alcohol use disorder, percentage who received brief counseling
Number of adults who received medication for substance use disorder | 12 months
  Of people aged 18 or older who screened positive for substance use disorder and/or alcohol use disorder, number who received medication
Number of adults who received medication for substance use disorder | 24 months
  Of people aged 18 or older who screened positive for substance use disorder and/or alcohol use disorder, number who received medication
Percentage of adults who received medication for substance use disorder | 24 months
  Of people aged 18 or older who screened positive for substance use disorder and/or alcohol use disorder, percentage who received medication
Percentage of adults who received medication for substance use disorder, including alcohol use disorder | 12 months
  Of people aged 18 or older who screened positive for substance use disorder and/or alcohol use disorder, percentage who received medication
Number of adults who received medication for substance use disorder, including alcohol use disorder, and adhered to 6 months of treatment | 12 months
  Of those aged 18 or older who received medication for substance use disorder and/or alcohol use disorder, number who adhered to treatment for 6 months
Number of adults who received medication for substance use disorder, including alcohol use disorder, and adhered to 6 months of treatment | 24 months
  Of those aged 18 or older who received medication for substance use disorder and/or alcohol use disorder, number who adhered to treatment for 6 months
Percentage of adults who received medication for substance use disorder, including alcohol use disorder, and adhered to 6 months of treatment | 24 months
  Of those aged 18 or older who received medication for substance use disorder and/or alcohol use disorder, percentage who adhered to treatment for 6 months
Percentage of adults who received medication for substance use disorder, including alcohol use disorder, and adhered to 6 months of treatment | 12 months
  Of those aged 18 or older who received medication for substance use disorder and/or alcohol use disorder, percentage who adhered to treatment for 6 months
Number of adults referred to specialty care for substance use disorder and/or alcohol use disorder | 12 months
  Of those aged 18 or older who were identified as having substance use disorder and/or alcohol use disorder, number who were referred to specialty care (psychiatry, 12-step programs, counseling, etc.)
Number of adults referred to specialty care for substance use disorder and/or alcohol use disorder | 24 months
  Of those aged 18 or older who were identified as having substance use disorder and/or alcohol use disorder, number who were referred to specialty care (psychiatry, 12-step programs, counseling, etc.)
Percentage of adults referred to specialty care for substance use disorder and/or alcohol use disorder | 24 months
  Of those aged 18 or older who were identified as having substance use disorder and/or alcohol use disorder, percentage who were referred to specialty care (psychiatry, 12-step programs, counseling, etc.)
Percentage of adults referred to specialty care for substance use disorder and/or alcohol use disorder | 12 months
  Of those aged 18 or older who were identified as having substance use disorder and/or alcohol use disorder, percentage who were referred to specialty care (psychiatry, 12-step programs, counseling, etc.)
Number of adults with alcohol use disorder | 12 months
  Of those aged 18 or older who were screened for substance use disorder, number who had alcohol use disorder
Number of adults with alcohol use disorder | 24 months
  Of those aged 18 or older who were screened for substance use disorder, number who had alcohol use disorder
Percentage of adults with alcohol use disorder | 24 months
  Of those aged 18 or older who were screened for substance use disorder, percentage who had alcohol use disorder
Percentage of adults with alcohol use disorder | 12 months
  Of those aged 18 or older who were screened for substance use disorder, percentage who had alcohol use disorder
Number of adults who received any evidence-based intervention for alcohol use disorder | 12 months
  Of those aged 18 or older identified as having alcohol use disorder, number who received any evidence-based intervention (brief counseling, medication, referral to specialty care)
Number of adults who received any evidence-based intervention for alcohol use disorder | 24 months
  Of those aged 18 or older identified as having alcohol use disorder, number who received any evidence-based intervention (brief counseling, medication, referral to specialty care)
Percentage of adults who received any evidence-based intervention for alcohol use disorder | 24 months
  Of those aged 18 or older identified as having alcohol use disorder, percentage who received any evidence-based intervention (brief counseling, medication, referral to specialty care)
Percentage of adults who received any evidence-based intervention for alcohol use disorder | 12 months
  Of those aged 18 or older identified as having alcohol use disorder, percentage who received any evidence-based intervention (brief counseling, medication, referral to specialty care)
Number of adults who received brief counseling for alcohol use disorder | 12 months
  Of those aged 18 or older identified as having alcohol use disorder, number who received brief counseling
Number of adults who received brief counseling for alcohol use disorder | 24 months
  Of those aged 18 or older identified as having alcohol use disorder, number who received brief counseling
Percentage of adults who received brief counseling for alcohol use disorder | 24 months
  Of those aged 18 or older identified as having alcohol use disorder, percentage who received brief counseling
Percentage of adults who received brief counseling for alcohol use disorder | 12 months
  Of those aged 18 or older identified as having alcohol use disorder, percentage who received brief counseling
Number of adults who received medication for alcohol use disorder | 12 months
  Of those aged 18 or older identified as having alcohol use disorder, number who received medication
Number of adults who received medication for alcohol use disorder | 24 months
  Of those aged 18 or older identified as having alcohol use disorder, number who received medication
Percentage of adults who received medication for alcohol use disorder | 24 months
  Of those aged 18 or older identified as having alcohol use disorder, percentage who received medication
Percentage of adults who received medication for alcohol use disorder | 12 months
  Of those aged 18 or older identified as having alcohol use disorder, percentage who received medication
Number of adults who received medication for alcohol use disorder and adhered to 6 months of treatment | 12 months
  Of those aged 18 or older who received medication for alcohol use disorder, number who adhered to treatment for 6 months
Number of adults who received medication for alcohol use disorder and adhered to 6 months of treatment | 24 months
  Of those aged 18 or older who received medication for alcohol use disorder, number who adhered to treatment for 6 months
Percentage of adults who received medication for alcohol use disorder and adhered to 6 months of treatment | 24 months
  Of those aged 18 or older who received medication for alcohol use disorder, percentage who adhered to treatment for 6 months
Percentage of adults who received medication for alcohol use disorder and adhered to 6 months of treatment | 12 months
  Of those aged 18 or older who received medication for alcohol use disorder, percentage who adhered to treatment for 6 months
Number of adults referred to specialty care for alcohol use disorder | 12 months
  Of those aged 18 or older who were identified as having alcohol use disorder, number who were referred to specialty care (psychiatry, 12-step programs, counseling, etc.)
Number of adults referred to specialty care for alcohol use disorder | 24 months
  Of those aged 18 or older who were identified as having alcohol use disorder, number who were referred to specialty care (psychiatry, 12-step programs, counseling, etc.)
Percentage of adults referred to specialty care for alcohol use disorder | 24 months
  Of those aged 18 or older who were identified as having alcohol use disorder, percentage who were referred to specialty care (psychiatry, 12-step programs, counseling, etc.)
Percentage of adults referred to specialty care for alcohol use disorder | 12 months
  Of those aged 18 or older who were identified as having alcohol use disorder, percentage who were referred to specialty care (psychiatry, 12-step programs, counseling, etc.)
Number of adults screened for substance use disorder | 24 months
  Number of people aged 18 and older who are screened for substance use disorder using a validated screening tool
Percent of adults screened for substance use disorder | 24 months
  Percent of people aged 18 and older who are screened for substance use disorder using a validated screening tool

OTHER OUTCOMES:
Association between implementation effectiveness and putative moderators and mediators | 12 months
  Longitudinal mixed-methods evaluation (surveys, interviews) to describe the association between implementation effectiveness and putative moderators (e.g., organizational readiness for change) and mediators (e.g., implementation climate)
Association between implementation effectiveness and putative moderators and mediators | 24 months
  Longitudinal mixed-methods evaluation (surveys, interviews) to describe the association between implementation effectiveness and putative moderators (e.g., organizational readiness for change) and mediators (e.g., implementation climate)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Jonas, MD, MPH, Principal Investigator — Ohio State University
Locations (3):
- United States (3):
  - Bon Secours Mercy Health, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Ohio Association of Community Health Centers, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jonas DE, Brill SB, Fried M, Brouwer L, Riley S, MacEwan SR, Hyer M, Palettas M, Hall OT, Vilensky M, Teater J, Carson WF 2nd, Wei L, Garner BR. The STop UNhealthy substance use now (STUN II) trial: protocol for a 48-site cluster randomized 2 x 2 factorial implementation trial to improve evidence-based screening and interventions for substance use disorder within primary care. Implement Sci. 2025 Sep 30;20(1):40. doi: 10.1186/s13012-025-01454-3. PMID 41029867